CLINICAL TRIAL: NCT03148171
Title: Project WERK (Wellness Encouragement Respect Kinship): Network Support to Engage and Retain Younger Black MSM in PrEP Care
Brief Title: Project WERK (Wellness Encouragement Respect Kinship)
Acronym: WERK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Howard Brown Health Center (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB17-0152; R34MH111392 (NIH)
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: HIV Prevention
Keywords: Pre-Exposure Prophylaxis (PrEP); Retention in PrEP Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Routine PrEP Care (No Intervention): Routine PrEP Care at each clinical site.
- WERK Supportive Contact (Active Comparator): Support contact will provide emotional support and practical support in order to help their friend/family member to stay engaged in PrEP Care.
  Interventions: Other: WERK Supportive Contact

INTERVENTIONS:
Other: WERK Supportive Contact — Provide emotional support and practical support. Support friend/family by helping him to stay engaged in PrEP Care.
  Arms: WERK Supportive Contact

SUMMARY:
The Project WERK intervention is a brief, theory based and culturally sensitive intervention designed to capitalize on organic yet underutilized social support networks in the lives of young black men who have sex with men (YBMSM). The intervention has been developed with input from clients and their support network members, case managers, social workers, primary care providers. The goal of the intervention is to improve retention in PrEP care for young Black MSM.

DETAILED DESCRIPTION:
Project WERK will recruit, consent and randomize 160 men, with 80 men randomized to each arm of the study. Men randomized to the control condition will receive standard PrEP care at each clinical site. Men randomized to the experimental condition will receive standard PrEP care and also will be asked to recruit a supportive contact from their social network. The support contact will then be engaged in a brief intervention designed to support their friend/family member around PrEP Care. Men and support contacts in the WERK intervention also will receive booster sessions via telephone and text. All participants will complete surveys at baseline and at three and twelve months post intervention.

ELIGIBILITY:
Inclusion criteria

Index subjects:

* Self-identify as African American/Black;
* Assigned male sex at birth;
* Any same gender anal or oral sex in the past 2 years;
* English speaking;
* Have at least one support contact in their network;
* Own a cell phone not shared with other persons;
* Between the ages of 18-35 years old; and
* Have had fewer than 3 PrEP clinical visits in the past 12 months.

Support Contact:

* Index participant has agreed to including the support contact
* Willing to attend face to face and telephone mini-booster sessions;
* 18 years of age or older;
* English speaking; and
* Owns a cell phone that is not shared with other persons.

Exclusion Criteria

Index Subject:

* Unable to provide informed consent;
* Plan to move out of the area within the next 12 months;
* Are not willing to attend intervention sessions; or
* Not willing to return for assessments.

For index participants without a support contact, we will refer them to an appropriate support group for PrEP.

Support Contact:

* Romantic partner of index participant;
* Unable to provide informed consent;
* Plan to move out of the area within the next 12 months;
* Are not willing to attend intervention sessions; or
* Not willing to return for assessments.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 290 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Retention in PrEP Care | 12-month
  Completing scheduled PrEP visits as determined by Electronic Medical Record (EMR) data

SECONDARY OUTCOMES:
HIV testing and STI testing | 12 months
  HIV serostatus and STI testing as determined by EMR data
Closeness and social support | 12 months
  Closeness and social support measures based on self-report

CONTACTS AND LOCATIONS:
Overall Officials: Alida Bouris, PhD, Principal Investigator — University of Chicago
Locations (1):
- Chicago Center for HIV Elimination, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No